CLINICAL TRIAL: NCT05402163
Title: Adaptive/Closed Loop vs. Continuous/Open Loop Deep Brain Stimulation of Subthalamic Nucleus: a Two-Phase, Cross-Over, Double-Blind Trial in Patients With Parkinson's Disease
Brief Title: CANadian Adaptive DBS TriAl
Acronym: CANADA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Alfonso Fasano, Professor - University of Toronto, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 17-5527
Record Dates: First submitted 2022-04-04; First posted 2022-06-02 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Continuous DBS (Other)
  Interventions: Device: Continuous DBS
- Adaptive DBS (Active Comparator)
  Interventions: Device: Adaptive DBS

INTERVENTIONS:
Device: Adaptive DBS — aDBS vs cDBS
  Arms: Adaptive DBS
Device: Continuous DBS — aDBS vs cDBS
  Arms: Continuous DBS

SUMMARY:
Parkinsonian symptoms, such as freezing of gait (FOG) or hypophonia, play a significant role in reducing quality of life for Parkinson disease (PD) patients, and are poorly responsive or can worsen with deep brain stimulation (DBS). Repeated adjustments of stimulation parameters may be beneficial however, continuous DBS (cDBS) does not adapt to the patients' rapidly fluctuating clinical status and does not take into account reliable and consistent state-trait biomarkers. These biomarkers can be recorded by the electrode itself as local field potentials (LFP). These LFPs can be used to guide stimulation output by means of a 'closed loop' or 'adaptive' DBS (aDBS).

This is a pilot, two-phase, double-blinded, cross-over study of chronic Adaptive vs. Continuous STN DBS in patients with PD by using a novel implantable DBS system that can automatically adjust stimulation parameters based on the patient's clinical condition. The study will test the hypothesis that aDBS stimulation will treat motor fluctuations similarly to continuous stimulation but it will be superior to the latter in the treatment of speech, gait impairment and falls.

ELIGIBILITY:
Inclusion Criteria:

* PD treated with bilateral STN DBS using Medtronic lead
* Able to provide informed consent and comply with study protocol
* Need to replace the implantable pulse generator (IPG) due to battery end of life
* Presence of disabling gait and/or balance and/or speech issues, as clinically judged by the PI and the patient
* Evidence that these disabling gait and/or balance and/or speech issues are worsened by DBS, i.e. they improve after turning DBS off.
* Use of contact 1 and/or 2 on one hemisphere and/or 9 and/or 10 on the other one
* Good LFP signal (assessable only after IPG replacement with Percept) in at least one hemisphere

Exclusion Criteria:

* Previous DBS surgery without Medtronic products
* Potential use of any therapeutic stimulation configuration (such as bipolar) during the study which will prevent the use of aDBS
* Presence of any other disorders potentially impacting the outcome measures (e.g. orthopaedic issues)
* Medically unstable
* Severe non-motor problems, such as depression, dementia, etc.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Activities of Daily Living using the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part II | Baseline, 5 months after IPG change, 8 months after battery change
  Unified Parkinson's Disease Rating Scale (MDS-UPDRS) II: Motor Aspects of Experiences of Daily Living (M-EDL), range 0-52. Lower scores reflect better motor experience.
Change in Quality of Life (QoL) using Parkinson's Disease Questionnaire (PDQ39) | Baseline, 5 months after IPG change, 8 months after battery change
  Parkinson's Disease Questionnaire (PDQ39): 8 dimensions, 5-point ordinal scoring system, each dimension total score range from 0 to 100. Lower scores reflect better QoL.
Change in Gait using the Zeno Walkway by Protokinetics | Baseline, 5 months after IPG change, 8 months after battery change
  Gait analysis (off and on medication) using the Zeno Walkway by Protokinetics.
Change in Speech Quality using the Praat software (Phonetic Sciences) | Baseline, 5 months after IPG change, 8 months after battery change
  Phonetic speech analysis (off and on medication) using the Praat software (Phonetic Sciences, Amsterdam, The Netherlands). Increased phonation reflects better speech quality.

SECONDARY OUTCOMES:
Change in Motor Outcomes (adaptive DBS vs continuous DBS arms) using Unified Parkinson's Disease Rating Scale part III (motor examination) | Baseline, 2-5 months after IPG change, 8 months after battery change
  Unified Parkinson's Disease Rating Scale motor examination (MDS-UPDRS III) score, range 0-132. Lower scores reflect less motor impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- Movement Disorders Centre - Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No